CLINICAL TRIAL: NCT00838773
Title: HIV Prevention Within High-Risk Social Networks
Brief Title: International Social Network Intervention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jeffrey Kelly, Professor of Psychiatry and Behavioral Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01DA023854 (NIH); 9R01DA023854 (NIH)
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- YMSM (Experimental): Young Men Who Have Sex with Men
  Interventions: Behavioral: YMSM
- YHA (Experimental): Young Heterosexual Adults
  Interventions: Behavioral: YHA
- ROMA (Experimental): Gypsies (Bulgarian)
  Interventions: Behavioral: ROMA
- Control (No Intervention): All study participants (including those in control condition networks) receive HIV/AIDS/STD risk reduction counseling at baseline, as well as testing and treatment or treatment referral for STDs and HIV infection. STD/HIV testing and treatment or treatment referral are provided at each followup point. This constitutes the control intervention.

INTERVENTIONS:
Behavioral: YMSM — Leaders of networks in the experimental condition will participate in a 9-session intervention training program that will inspire and assist leaders to communicate HIV prevention risk reduction messages with their immediate friends. The first five sessions will focus on HIV risk predictors including HIV/AIDS knowledge, safer sex peer norms, condom attitudes, condom use intentions, and self-efficacy in remaining safe. The remaining four sessions will reinforce the leaders for continuing their HIV prevention communications and remind them of the topics during the main sessions.
  Arms: YMSM
Behavioral: YHA — Leaders of networks in the experimental condition will participate in a 9-session intervention training program that will inspire and assist leaders to communicate HIV prevention risk reduction messages with their immediate friends. The first five sessions will focus on HIV risk predictors including HIV/AIDS knowledge, safer sex peer norms, condom attitudes, condom use intentions, and self-efficacy in remaining safe. The remaining four sessions will reinforce the leaders for continuing their HIV prevention communications and remind them of the topics during the main sessions.
  Arms: YHA
Behavioral: ROMA — Leaders of networks in the experimental condition will participate in a 9-session intervention training program that will inspire and assist leaders to communicate HIV prevention risk reduction messages with their immediate friends. The first five sessions will focus on HIV risk predictors including HIV/AIDS knowledge, safer sex peer norms, condom attitudes, condom use intentions, and self-efficacy in remaining safe. The remaining four sessions will reinforce the leaders for continuing their HIV prevention communications and remind them of the topics during the main sessions.
  Arms: ROMA

SUMMARY:
This grant involves 24 social networks of young men who have sex with men, Roma, and young high-risk heterosexual adult men and women living in Hungary, Bulgaria and Russia.

DETAILED DESCRIPTION:
For over 4 years, our international collaborative research team has carried out a social network HIV prevention intervention trial with community populations of young men who have sex with men (YMSM), disadvantaged ethnic minority Roma (Gypsies), and high-risk heterosexual adult (YHA) women and men in Hungary, Bulgaria and Russia. Eastern Europe has seen a sharp increase in HIV incidence, and social network interventions are high in cultural relevance because post-communist populations have a long history of trusting and relying upon their personal networks more than their governments. Across the three countries represented in our research during the past funding period, we enrolled social networks of YMSM, Roma, and YHAs. This study will renew our international collaboration to extend this network intervention approach. Our study, to date, has worked with very small independent friendship groups (usually composed of 5-6 people) as "egocentric" social networks.

ELIGIBILITY:
Inclusion Criteria:Members of a friendship group will be eligible for enrollment if they are of legal age to independently consent to participate in this study. In its review and approval of this protocol, the IRB at BotkinHospital, St. Petersburg, Russia verified and confirmed in writing to us that the age of research participation consent is 15. In its review and approval of this protocol, the IRB at the Health and Social Development Foundation determined that the age of research participation consent in Bulgaria is 16. In Hungary, the IRB at the Institute of Sociology at the Hungarian Academy of Sciences determined that the age of independent consent to participate in this study is 14.

-

Exclusion Criteria:Individuals will be excluded from enrollment into the study if they are below the age for providing independent consent or are not capable of providing informed consent based on impairment due to the presence of sever psychopatology, substance use, or similar conditions observed at the time of informed consent. Social networks will be excluded from the study if: (1) more than 33% of named network members do not agree to participate; (2) fewer than 50% of members report occurrence of unprotected intercourse during the past 3 months at baseline; or (3) more than 10% of a network's members are also members of another network enrolled in the study.

-

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1292 (Actual)
Dates: Start 2007-05; Primary Completion 2012-04 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Target effect of at least 30% consistent condom use among the experimental intervention group at 15-month followup. | August 2015

SECONDARY OUTCOMES:
15-month cumulative STD incidence rate of 20% among the control group compared 10% or less among the experimental group. | August 2015

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey A, Kelly, PhD, Principal Investigator — Medical College of Wisconsin; Yuri A. Amirkhanian, Ph.D., Study Director — Medical College of Wisconsin; Judit Takacs, Ph.D., Study Director — Institute of Sociology of Hungarian Academy of Sciences; Elena Kabakchieva, MD, Study Director — Health and Social Development Foundation
Locations (3):
- Health and Social Development Foundation, Sofia, Bulgaria
- Hungarian Academy of Sciences, Budapest, Hungary
- Botkin Hospital for Infectious Diseases #30, Saint Petersburg, Russia

REFERENCES:
- [Result] Takacs J, Kelly JA, P Toth T, Mocsonaki L, Amirkhanian YA. Effects of Stigmatization on Gay Men Living with HIV/AIDS in a Central-Eastern European Context: A Qualitative Analysis from Hungary. Sex Res Social Policy. 2013 Mar 1;10(1):24-34. doi: 10.1007/s13178-012-0102-5. Epub 2012 Oct 25. PMID 23439743
- [Result] Amirkhanian YA. Social networks, sexual networks and HIV risk in men who have sex with men. Curr HIV/AIDS Rep. 2014 Mar;11(1):81-92. doi: 10.1007/s11904-013-0194-4. PMID 24384832
- [Result] Amirkhanian YA, Kelly JA, Takacs J, McAuliffe TL, Kuznetsova AV, Toth TP, Mocsonaki L, DiFranceisco WJ, Meylakhs A. Effects of a social network HIV/STD prevention intervention for MSM in Russia and Hungary: a randomized controlled trial. AIDS. 2015 Mar 13;29(5):583-93. doi: 10.1097/QAD.0000000000000558. PMID 25565495
- [Result] Amirkhanian YA, Kelly JA, Kabakchieva E, Antonova R, Vassileva S, Difranceisco WJ, McAuliffe TL, Vassilev B, Petrova E, Khoursine RA. High-risk sexual behavior, HIV/STD prevalence, and risk predictors in the social networks of young Roma (Gypsy) men in Bulgaria. J Immigr Minor Health. 2013 Feb;15(1):172-81. doi: 10.1007/s10903-012-9596-4. PMID 22370730